CLINICAL TRIAL: NCT04428398
Title: Urinary T Lymphocytes Predict Renal Flares in Patients With Inactive Anti-neutrophil Cytoplasmic Antibody (ANCA) Associated Glomerulonephritis
Brief Title: Urinary T Lymphocytes Predict Renal Flares in Patients With Inactive ANCA-associated Glomerulonephritis
Acronym: PRE-FLARED
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Enghard, PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: PRE-FLARED
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Glomerulonephritis Acute
Keywords: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Pauci-Immune Glomerulonephritis; urinary biomarker; Churg-Strauss Syndrome; Microscopic Polyangiitis; Granulomatosis with Polyangiitis; effector memory T lymphocytes; prediction
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Churg-Strauss Syndrome; Microscopic Polyangiitis; Granulomatosis with Polyangiitis | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples (approximately 60 mL per patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No renal involvement: Patients with ANCA-vasculitis and no ANCA-associated renal involvement in disease history
  Interventions: Diagnostic Test: Analysis of urine samples with flow cytometry
- Renal remission: Patient with ANCA-vasculitis in renal remission
  Interventions: Diagnostic Test: Analysis of urine samples with flow cytometry

INTERVENTIONS:
Diagnostic Test: Analysis of urine samples with flow cytometry — Urine samples will be conserved and frozen upon arrival. All samples will be stained according to T cell and TEC (tubular epithelial cells) panel with fluorochromes.
  T cell panel: CD3, CD4, CD8, CCR7, CD45RO, CD28, CD279; TEC panel: vimentin, cytokeratine, CD10, CD13, CD227, CD326

SUMMARY:
Urinary CD4+ and CD8+ T lymphocytes may predict renal flares in patients with inactive ANCA-associated vasculitis and thus serve as early non-invasive biomarkers. Urine samples of patients with inactive renal ANCA-vasculitis will be analysed by flow cytometry and compared to clinical outcome after 6 months.

DETAILED DESCRIPTION:
Data of previous studies have shown that counts of urinary T lymphocyte subsets correlate with disease activity in several immunological renal diseases, e.g. ANCA-associated glomerulonephritis. Thus, study authors hypothesise that CD4+, respectively CD8+, T effector memory lymphocytes found in urine samples of patients with inactive ANCA-vasculitis predict subsequent renal flares. Therefore, quantification of these cellular subsets might reliably predict relapse of ANCA associated glomerulonephritis at an early stage. In a prospective experimental study urine of patients with ANCA-vasculitis and no renal involvement or patients in renal remission will be analysed by flow cytometry. After 6 months of observation, clinical outcome and potential renal relapse will be determined and correlated to initial T lymphocyte count.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed ANCA-associated vasculitis (clinical diagnosis of granulomatosis with polyangiitis, eosinophilic granulomatosis with polyangiitis or microscopic polyangiitis consistent with the Chapel-Hill consensus definitions AND positive test for proteinase 3-ANCA or myeloperoxidase-ANCA)
* no currently active renal involvement (defined as BVAS = 0 with exception of hematuria or proteinuria as signs of renal scars)
* written and informed consent

Exclusion Criteria:

* urinary tract infection
* active menstrual bleeding
* active renal involvement
* other active renal disease (e.g. diabetic nephropathy)

Initially, we defined treatment with rituximab as exclusion criteria. However, upon closer examination, we recognized that this exclusion criterion was overly restrictive and may have inadvertently excluded eligible participants who met our other inclusion criteria. As a result of this reassessment, we have revised our exclusion criteria to no longer exclude individuals solely on the basis of receiving rituximab treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in medical wards or at outpatient departments of 2 facilities:
  * Charité - Universitätsmedizin Berlin
  * Helios Klinikum Berlin-Buch
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Prediction of renal relapse after six months depending initial CD4+ count | 6 months
  * relapse defined as Birmingham Vasculitis Activity Score (BVAS) > 1 + at least one renal element or
  * intensified treatment regime (Prednisolon equivalent > 20 mg/d or novel induction treatment with Rituximab or Cyclophosphamide)

SECONDARY OUTCOMES:
Prediction of renal relapse after six months depending initial CD8+ count | 6 months
Prediction of renal relapse after six months depending initial CD4+/CD8+ subsets | 6 months
  Subsets: T effector memory cells (CD45RO+/CCR7-)
Prediction of renal relapse after 12 months depending initial CD4+ count | 12 months
Prediction of renal relapse after 12 months depending initial CD8+ count | 12 months
Prediction of renal relapse after 12 months depending initial CD4+/CD8+ subsets | 12 months
  Subsets: T effector memory cells (CD45RO+/CCR7-)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Enghard, Principal Investigator — Charite University, Berlin, Germany; Adrian Schreiber, PD Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Helios Klinikum Berlin-Buch, Berlin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Goceroglu A, Berden AE, Fiocco M, Flossmann O, Westman KW, Ferrario F, Gaskin G, Pusey CD, Hagen EC, Noel LH, Rasmussen N, Waldherr R, Walsh M, Bruijn JA, Jayne DR, Bajema IM; European Vasculitis Society (EUVAS). ANCA-Associated Glomerulonephritis: Risk Factors for Renal Relapse. PLoS One. 2016 Dec 14;11(12):e0165402. doi: 10.1371/journal.pone.0165402. eCollection 2016. PMID 27973575
- [Background] Menez S, Hruskova Z, Scott J, Cormican S, Chen M, Salama AD, Alasfar S, Little MA, Safrankova H, Honsova E, Tesar V, Geetha D. Predictors of Renal Outcomes in Sclerotic Class Anti-Neutrophil Cytoplasmic Antibody Glomerulonephritis. Am J Nephrol. 2018;48(6):465-471. doi: 10.1159/000494840. Epub 2018 Nov 23. PMID 30472700
- [Background] Cordova-Sanchez BM, Mejia-Vilet JM, Morales-Buenrostro LE, Loyola-Rodriguez G, Uribe-Uribe NO, Correa-Rotter R. Clinical presentation and outcome prediction of clinical, serological, and histopathological classification schemes in ANCA-associated vasculitis with renal involvement. Clin Rheumatol. 2016 Jul;35(7):1805-16. doi: 10.1007/s10067-016-3195-z. Epub 2016 Feb 6. PMID 26852317
- [Background] Enghard P, Rieder C, Kopetschke K, Klocke JR, Undeutsch R, Biesen R, Dragun D, Gollasch M, Schneider U, Aupperle K, Humrich JY, Hiepe F, Backhaus M, Radbruch AH, Burmester GR, Riemekasten G. Urinary CD4 T cells identify SLE patients with proliferative lupus nephritis and can be used to monitor treatment response. Ann Rheum Dis. 2014 Jan;73(1):277-83. doi: 10.1136/annrheumdis-2012-202784. Epub 2013 Mar 8. PMID 23475982
- [Background] Abdulahad WH, Kallenberg CG, Limburg PC, Stegeman CA. Urinary CD4+ effector memory T cells reflect renal disease activity in antineutrophil cytoplasmic antibody-associated vasculitis. Arthritis Rheum. 2009 Sep;60(9):2830-8. doi: 10.1002/art.24747. PMID 19714581
- [Derived] Prskalo L, Skopnik CM, Goerlich N, Freund P, Wagner L, Grothgar E, Mirkheshti P, Klocke J, Sonnemann J, Metzke D, Schneider U, Hiepe F, Eckardt KU, Salama AD, Bieringer M, Schreiber A, Enghard P. Urinary CD4 + T Cells Predict Renal Relapse in ANCA-Associated Vasculitis. J Am Soc Nephrol. 2024 Apr 1;35(4):483-494. doi: 10.1681/ASN.0000000000000311. Epub 2024 Jan 17. PMID 38231590